CLINICAL TRIAL: NCT05100992
Title: Prospective Global Registry of Percutaneous Coronary Intervention in Bifurcation Lesions (PROGRESS-BIFURCATION)
Brief Title: Progress Bifurcation Global Registry
Status: Recruiting | Type: Observational
Sponsor: Minneapolis Heart Institute Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: PROGRESS-BIFURCATION
Record Dates: First submitted 2021-09-20; First posted 2021-10-29 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Coronary Artery Disease; Coronary Bifurcation Lesions
Keywords: bifurcation lesions; percutaneous coronary intervention
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Percutaneous Coronary Interbention — Percutaneous Coronary Interbention

SUMMARY:
Coronary bifurcation lesions are lesions (or blockages) that occur at or near the intersection of a major coronary artery and one of the arteries' side branches.

Numerous techniques and devices have been developed to treat coronary bifurcations; however, these types of lesions remain some of the most challenging, both in terms of procedural success and outcome. This study is designed as an observational, multi-center registry that will collect information on treatment strategies and outcomes of consecutive patients undergoing percutaneous coronary interventions (PCI) in coronary bifurcations among various participating centers, in order to determine the frequency of bifurcation PCI, the procedural strategies utilized, and the procedural outcomes.

DETAILED DESCRIPTION:
Numerous techniques and devices have been developed to treat coronary bifurcations; however, these types of lesions remain some of the most challenging, both in terms of procedural success and outcome. Several techniques are currently being utilized to treat coronary bifurcation lesions, including a 1-stent provisional stenting technique. Various 2-stent techniques are also performed, including: double kiss crush (DK crush4), culotte, T and protrusion (TAP), crush, mini-crush, reverse crush and V-stenting. The optimal technique for bifurcation stenting when two stents are required remains controversial; however, the DK crush technique appears to have stronger data, especially for left main bifurcations. However, DK crush can be challenging to perform, requiring several steps and frequent troubleshooting.

The adoption of DK crush and other 2-stent bifurcation strategies, as well as the rigor of implementation, have received limited study. This study is designed as an observational, multi-center registry that will collect information on treatment strategies and outcomes of consecutive patients undergoing percutaneous coronary interventions (PCI) in coronary bifurcations among various participating centers, in order to determine the frequency of bifurcation PCI, the procedural strategies utilized,

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* undergoing bifurcation percutaneous coronary intervention

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects over 18 years of age and undergoing bifurcation percutaneous coronary intervention at each of the participating center.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2020-04-23 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Procedural Success During Bifurcation PCI | From Date of Procedure to Date of Hospital Discharge, approximately 48-72 hrs after index procedure.
  procedural success is defined as the absence of in-hospital major cardiac adverse events (MACE), including any of the following adverse events prior to hospital discharge: death, stroke, myocardial infarction, recurrent angina requiring urgent repeat target vessel revascularization with PCI or coronary bypass surgery, and tamponade requiring pericardiocentesis or surgery.

SECONDARY OUTCOMES:
Technical Success | From Date of Procedure to Date of Hospital Discharge, approximately 48-72 hrs after index procedure.
  Technical success will be defined as successful bifurcation lesion recanalization by any method with achievement of < 30% residual stenosis and TIMI 3 flow in both the main vessel and side branch.

CONTACTS AND LOCATIONS:
Locations (1):
- Minneapolis Heart Institute Foundation, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Strepkos D, Alexandrou M, Mutlu D, Carvalho PEP, Ser OS, Jalli S, Voudris K, Burke MN, Sandoval Y, Brilakis ES. Impact of Side Branch Occlusion on Patient Outcomes After Bifurcation Percutaneous Coronary Intervention. Catheter Cardiovasc Interv. 2025 Apr;105(5):1142-1148. doi: 10.1002/ccd.31439. Epub 2025 Feb 3. PMID 39898485
- [Derived] Simsek B, Kostantinis S, Karacsonyi J, Allana S, Vemmou E, Nikolakopoulos I, Burke MN, Garcia S, Wang Y, Chavez I, Gossl M, Sorajja P, Mooney M, Poulose A, Sandoval Y, Traverse J, Rangan BV, Brilakis ES. Outcomes and challenges of the provisional stenting technique: Insights from the PROGRESS-BIFURCATION registry. Catheter Cardiovasc Interv. 2022 Nov;100(5):749-755. doi: 10.1002/ccd.30401. Epub 2022 Sep 19. PMID 36121014
- [Derived] Simsek B, Kostantinis S, Karacsonyi J, Vemmou E, Nikolakopoulos I, Assali M, Burke MN, Garcia S, Wang Y, Chavez I, Goessl M, Sorajja P, Mooney M, Poulose A, Traverse J, Rangan BV, Brilakis ES. Challenges and outcomes of the double kissing crush stenting technique: Insights from the PROGRESS-BIFURCATION registry. Catheter Cardiovasc Interv. 2022 Mar;99(4):1038-1044. doi: 10.1002/ccd.30135. Epub 2022 Feb 23. PMID 35195331